CLINICAL TRIAL: NCT04978168
Title: Using Implementation Interventions and Peer Recovery Support to Improve Opioid Treatment Outcomes in Community Supervision
Brief Title: Opioid Treatment and Peer Recovery Support
Acronym: JCOIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Temple University (Other); University of Rhode Island (Other); The Miriam Hospital (Other); National Institute on Drug Abuse (NIDA) (NIH); CODAC Behavioral Healthcare (Unknown); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2002002636; U01DA050442-01 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-07-27 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Opioid-use Disorder
Keywords: Opioid Use; Medications for Opioid Use
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A Type 1 hybrid implementation-effectiveness study conducted in two phases. The first recruits as staff/leaders from probation agencies and community treatment agencies. The second phase (which starts after the implementation in the first period is completed) recruits adults on probation and staff of probation agencies. The Core Implementation study (first phase) involves a pre-post design. The effectiveness study (second phase) uses randomized parallel assignment with two arms.
  The initial Core Implementation study involved four phases: Exploration (baseline), Preparation, Implementation, Sustainability (6- and 12-month follow-ups). The subsequent Effectiveness study starts after the Implementation phase is completed, with its own baseline data and follow-ups up to 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Implementation Core (Experimental): During baseline Exploration, staff organizational surveys are collected. During Preparation, staff focus groups conduct needs assessment with system mapping of linkage points for screening, assessment, and referral, and the agencies/staff involved in these activities. During Implementation, sites use facilitated local change teams (LCT) provided with a core set implementation strategies to facilitate linkages between probation agencies and local community treatment providers. The LCTs identify barriers to change, approaches to overcome barriers, do goal selection using SMART (specific, measurable, achievable, relevant, timely) goals and evidence for medications, address stigma, and clarify needs/expectations/roles of probation officers and treatment providers, then choose and implement goals and strategies. Sustainability Phase: Facilitators work with LCTs for 12 months using a written action plan based on goal selection.
  Interventions: Behavioral: Core Intervention
- Randomized Trial of Peer Support Specialist Model (Experimental): After Core implementation is complete, half of adult participants in probation who consent will be randomly assigned to a Peer Support Specialist (PSS) condition. PSS are assigned to adults diagnosed with OUD within 6 months of entry into probation, in addition to treatment as usual. PSS establish linkages to community providers (medical, mental health, substance use treatment); educate about recovery support services, transportation assistance, MOUD; provide experiential, non-clinical support to individuals with SUD; share skills, offer support for setting goals and navigating the recovery process); and provide referrals and support for treatment, housing, employment, drug court, and probation.
  Interventions: Behavioral: Peer Support Specialists (PSS)
- Randomized to Treatment as Usual (Active Comparator): After Core Implementation is complete, half of adult participants in probation who consent will be randomly assigned to continue with usual care.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Core Intervention — Staff are provided with a core set of implementation strategies to facilitate interorganizational linkages between probation agencies and local community treatment providers.
  Arms: Implementation Core
Behavioral: Peer Support Specialists (PSS) — Participants randomized to PSS will meet with a PSS for 6 months. Contact scheduled is flexible and based on the participant's needs and wants, plus written guidance for PSS-participant interactions.
  Arms: Randomized Trial of Peer Support Specialist Model
Behavioral: Treatment as Usual (TAU) — Participants randomized to TAU will receive the services that will be offered at the time the Core Implementation intervention is completed.
  Arms: Randomized to Treatment as Usual

SUMMARY:
Determine whether a facilitated local change team intervention improves a probation organization's client-level medication for opioid use disorder (MOUD) outcomes and implementation outcomes relative to baseline across multiple sites. Determine whether client-level outcomes are further enhanced by the introduction of Peer Support Services.

DETAILED DESCRIPTION:
Background: The purpose is to determine whether a facilitated local change team (LCT) intervention improves linkage to medication for opioid use disorder (MOUD) and implementation outcomes, and whether participant-level outcomes are further enhanced by the use of Peer Support Specialists (PSS).

Methods/Design: This Type 1 hybrid implementation-effectiveness study involves a pre-post design (implementation study) followed by a randomized trail of PSS (effectiveness study). The study is conducted at 7 performance sites in 3 states.

Phase 1 (Core Implementation Study): The Exploration, Preparation, Implementation, Sustainability (EPIS) framework is used to guide system-change through facilitated LCTs consisting of probation and community treatment staff who are given a core set of implementation strategies which are used to conduct a needs assessment and set goals. The overall objective is to improve linkage to the continuum of evidence-based care for justice-involved individuals with opioid use disorder (OUD). Organizational (program-level) and staff survey are collected at the end of each EPIS stage (baseline Exploration, end of Preparation, end of Implementation, and 12 months [Sustainability]). Implementation outcomes: Organizational engagement in MOUD (primary), plus changes in staff knowledge/attitudes and organizational outcomes (secondary).

Phase 2 (Effectiveness Study of PSS): After completing implementation, 450 adults on probation are randomized to receive PSS vs. treatment as usual (TAU), with assessments at baseline, 3, and 6 months. This trial tests whether having a trained peer improves clinical outcomes beyond effects of Core Implementation. Implementation program-level outcomes include organizational engagement in MOUD use (primary outcome); changes in staff knowledge and attitudes about MOUD, commitment and efficacy, readiness for change; organizational attitudes for change, commitment and efficacy (secondary outcomes). Client-level effectiveness outcomes include participant engagement in MOUD (primary outcome), probation revocation, illicit opioid use, and overdoses (secondary outcomes). Other aims include identifying barriers and facilitators, and cost-benefit analysis of PSS.

Primary Research Questions:

The primary aim is to test the effectiveness of PSS compared to TAU (agency approach after implementation) on outcomes of individuals on probation: Engagement in MOUD (primary effectiveness outcome), probation revocation (secondary), illicit opioid use (secondary), and overdose (tertiary).

The second aim is to test the effectiveness of EPIS-based Core Implementation Intervention relative to baseline on engagement in MOUD (primary implementation outcome).

The third aim is to test the effects of the EPIS implementation strategies relative to baseline on program-level (organizational and staff-level) outcomes.

The fourth aim is to conduct a cost-benefit analysis of implementing PSS compared to TAU.

The fifth aim is to identify organizational and staff barriers and facilitators to intervention implementation by conducting qualitative interviews with key probation and community treatment stakeholders who are managing and delivering the MOUD program.

ELIGIBILITY:
Inclusion Criteria:

* Community Provider Staff: Any front-line treatment provider at an agency participating in this study who: (a) provides support to MOUD clients, (b) has an active caseload including some individuals on probation, and (c) willing to commit to 12 months to the project.
* Probation/Parole Staff: Any probation officer (PO) at an agency participating in this study who (a) has an active caseload, and (b) is willing to commit to 12 months to the project.
* Individuals on Probation: (a) 18 years or older, (b) committed to probation within 90 days prior to study enrollment, (c) English speaking, (d) diagnosed with OUD, (e) have stable method of contact in community

Exclusion Criteria:

* Individuals on Probation: Currently incarcerated or in a court-mandated inpatient treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Individual-Level Experimental (Period 2) Outcome: Engagement in MOUD | 26 weeks
  Calculated from self-report survey of being enrolled in MOUD (yes or no) at each assessment.
Program-Level Implementation Outcome: Engagement in MOUD | 26 weeks
  MOUD engagement (primary implementation outcome) is defined as enrollment in MOUD treatment program, or filling a prescription for buprenorphine from a provider (in not on MOUD at time of recruitment), or remaining in MOUD treatment (if already on MOUD when recruited or at previous follow-up), coded dichotomously. Number of clients in probation enrolled in MOUD is tracked via medical and probation records.

SECONDARY OUTCOMES:
Detainment during Assessment Period (Individual-Level Experimental (Period 2) Outcome) | 26 weeks
  Calculated from probation records: Number of days detained during the assessment period
Opioid Use (Individual-Level Experimental (Period 2) Outcome) | 26 weeks
  Calculated from self-report surveys and urine screens: any opioid use
Non-Fatal Overdose Events (Individual-Level Experimental (Period 2) Outcome) | 26 weeks
  Calculated from treatment agency records: number of reports of medical treatment or death due to overdose events.
Staff MOUD Knowledge and Attitudes (Program-Level Implementation Outcome) | 26 weeks
  Extent of staff knowledge about and attitudes towards MOUD, commitment and efficacy, readiness for change, using Medications Opinion Survey.
Organizational Readiness for Change (Program-Level Implementation Outcome) | 26 weeks
  Measures of organizational climate, functioning, innovation support, leadership, and staff attributes were adapted from the Evidence-Based Practices Attitudes Scale (Aarons, 2004), Survey of Organizational Functioning (IBR, 2005), and Organizational Readiness for Change (IBR, 2009). Organizational linkages for collaboration and coordination between correctional and treatment agency dyads, using the Inter-Organizational Relationships (IOR) Survey.
Input Costs: PSS time (Program-Level Implementation Outcome) | 26 weeks
  PSS logs will be used to record the time PSSs spend with each participant (hours and minutes). Data analyses will convert these to dollar costs per participant using information from the Bureau of Labor Statistics.
Input Costs: Medical Usage (Program-Level Implementation Outcome) | 26 weeks
  Participant surveys will be sued to record number of visits to each type of medical provider during the study. Data analyses will convert these to dollar costs using Medicare fee-for-service information.
Outcome Costs (Program-Level Implementation Outcome) | 26 weeks
  Participant surveys will be used to record number of days in jail during the follow-up period. Analyses will convert these to dollar costs using government information.

CONTACTS AND LOCATIONS:
Overall Officials: Rosemarie A Martin, PhD, Principal Investigator — Brown University; Damaris J Rohsenow, PhD, Principal Investigator — Brown University; Lauren Brinkley-Rubinstein, PhD, Principal Investigator — Duke University; Steven Belenko, PhD, Principal Investigator — Temple University; Lynda Stein, PhD, Principal Investigator — University of Rhode Island; Josiah Rich, MD, Principal Investigator — The Miriam Hospital
Locations (3):
- United States (3):
  - Duke University, Durham, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
The coordinating center is charged with creating de-identified versions of agency staff and probation individual level data available at the end of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after the results of the primary study analyses have been accepted for publication. The data will be available for five years.
Access Criteria: De-identified data will be shared with the Methodology and Advanced Analytics Resource Center (MAARC) of JCOIN and with qualified researchers on request to the MAARC.